CLINICAL TRIAL: NCT04306692
Title: Myo-inositol Versus Clomiphene Citrate as First Line Treatment for Ovulation Induction in PCOS
Brief Title: Myo-inositol Versus Clomiphene Citrate in PCOS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: clomiphene citrate is no longer being considered as standard treatment for polycystic ovary syndrome
Sponsor: University Hospital, Ghent (Other)
Collaborators: Gedeon Richter Plc. (Industry); University Hospital, Antwerp (Other); AZ Jan Palfijn Gent (Other); Our Lady of Lourdes Hospital Waregem (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004604-20
Record Dates: First submitted 2020-02-12; First posted 2020-03-13 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Ovulation Induction; Polycystic Ovary Syndrome; Clomiphene; Inositol
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol; Clomiphene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inositol group (Experimental): Myo-inositol 4000 mg Dosing: 2 x 1 bag per day, per os (subjects can take myo-inositol during the meal but it is not obliged) during 3 consecutive treatment cycles.
  Interventions: Drug: Myo-inositol
- Clomiphene citrate group (Active Comparator): Each tablet contains 50 mg of clomiphene citrate Dosing: 1 tablet per day, per os, from cycle day 3 until 7 (extremes included), stepping up until a maximum dose of 3 tablets per day for 5 consecutive days during 3 consecutive treatment cycles.
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Myo-inositol — 2 x 1 bag per day, per os (subjects can take myo-inositol during the meal but it is not obliged).
  Arms: Inositol group
Drug: Clomiphene Citrate — Each tablet contains 50 mg of clomiphene citrate which means 33,9 mg of clomiphene. Other constituents are sucrose, lactose monohydrate, corn starch, pregelatinized starch, yellow iron oxide (E172) and magnesium stearate (E470b).
  Dosing: 1 tablet per day from cycle day 3 until 7 (extremes included), stepping up until a maximum dose of 3 tablets per day for 5 consecutive days.
  Arms: Clomiphene citrate group

SUMMARY:
Specific aim: To compare inositol and the golden standard first line treatment of ovulation induction, namely clomiphene citrate.

ELIGIBILITY:
Inclusion Criteria:

* Rotterdam criteria for PCOS (cf. the recent ESHRE guidelines): at least 2 out of 3 criteria should be fulfilled: irregular cycle (shorter than 21 days or longer than 35 days); clinical (modified Ferriman-Gallwey score ≥ 6) or biochemical signs (elevated free testosterone) of hyperandrogenism (www.eshre.eu/Guidelines-and- Legal/Guidelines/Polycystic-Ovary-Syndrome.aspx); PCO ovaries on ultrasound (www.eshre.eu/Guidelines-and- Legal/Guidelines/Polycystic-Ovary-Syndrome.aspx): multiple small cysts (≥ 20 per ovary and/or an ovarian volume ≥ 10 ml, measured with a probe >8 MHz) in both ovaries.
* A first treatment cycle, possibly combined with intra uterine insemination (IUI) and this for (one of) the following reasons: mild male factor (as defined by each local center) endometriosis AFS score 1 or 2
* Use of own or donor sperm.

Exclusion Criteria:

* Tubal factors
* Uterine factors
* Endometriosis AFS score 3 or 4
* Moderate to severe male factor (as defined by each local center)
* BMI > 35

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of cumulative ongoing pregnancy (a pregnancy diagnosed by ultrasonic visualisation of one or more gestational sacs with fetal heart beat) after 3 treatment cycles with inositol versus clomiphene citrate for ovulation induction. | At 7 - 8 gestational weeks
  Recently, a meta-analysis on the use of inositol in PCOS was published. This study showed that inositol leads to a more regular menstrual cycle and recovery of ovarian function. Less data are present on pregnancy rates. No RCT was found on the comparison between inositol and the golden standard first line treatment of ovulation induction, namely clomiphene citrate. Another advantage of inositol is that it doesn't have side effects compared to metformin and that there is no elevated risk on multiple pregnancies, which is the case with clomiphene citrate.

SECONDARY OUTCOMES:
The number of potential adverse events | During 3 consecutive treatment cycles (each treatment cycle is up to 5 weeks)
  The potential adverse events will be measured to determine whether the compliance for the patient is acceptable.
The occurrence of ovulation | During 3 consecutive treatment cycles (each treatment cycle is up to 5 weeks)
  The occurence of ovulation will be measured to determine whether the compliance for the patient is acceptable.
The number of cancelled treatment cycles | During 3 consecutive treatment cycles (each treatment cycle is up to 5 weeks)
  The number of cancelled treatment cycles will be measured to determine whether the compliance for the patient is acceptable.
The number of multiple pregnancies | During 3 consecutive treatment cycles (each treatment cycle is up to 5 weeks)
  The number of multiple pregnancies will be measured to determine whether the compliance for the patient is acceptable.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent, Belgium